CLINICAL TRIAL: NCT03024112
Title: Impact of Prophylactic High Flow Nasal Oxygen in Post-Operative Thoracic Surgical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12-1403
Record Dates: First submitted 2017-01-10; First posted 2017-01-18 (Estimated); Results first posted 2017-12-05 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Post-operative Pulmonary Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Heated humidified high-flow nasal cannula (HHFNC) oxygen (Experimental): The intervention group received HHFNC O2 at a set flow of 40L/min. FiO2 was titrated by respiratory therapists to maintain SpO2 ≥ 90%. The HHFNC O2 apparatus included: 1) Air-Oxygen blender - capable of delivering 21-100% FiO2 at flow rates up to 60L/min, 2) Heated Humidifier - providing active heating and humidification to the delivered air-O2 blend, 3) Nasal cannula - larger diameter, slightly elongated nasal cannula with single limb connection to humidifier
  Interventions: Device: Heated humified high-flow nasal cannula Oxygen
- Standard oxygen Therapy (Active Comparator): The standard O2 treatment group received usual nasal cannula or face mask oxygen titrated by nurses as necessary to maintain SpO2 ≥ 90%.
  Interventions: Other: Standard oxygen therapy

INTERVENTIONS:
Device: Heated humified high-flow nasal cannula Oxygen
  Arms: Heated humidified high-flow nasal cannula (HHFNC) oxygen
Other: Standard oxygen therapy
  Arms: Standard oxygen Therapy

SUMMARY:
The Investigators goal was to study the effect of high flow nasal cannula oxygen (HFNC) on the rate of post-operative pulmonary complications in thoracic surgical patients. The Investigators hypothesis is that prophylactic HFNC oxygen, as compared to standard oxygen treatment, will reduce the incidence of postoperative pulmonary complications, improve post-operative pulmonary function, and reduce Intensive Care Unit (ICU) and hospital length of stay.

DETAILED DESCRIPTION:
The Investigators goal was to study the effect of high flow nasal cannula oxygen (HFNC) on the rate of post-operative pulmonary complications in thoracic surgical patients. The Investigators hypothesis is that prophylactic HFNC oxygen, as compared to standard oxygen treatment, will reduce the incidence of postoperative pulmonary complications, improve post-operative pulmonary function, and reduce ICU and hospital length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing Thoracic surgery
* Planned admission to ICU after surgery

Exclusion Criteria:

* Younger than 18
* Pregnant
* Breast feeding
* Known diagnosis of obstructive sleep apnea
* Current or previous lung transplant
* Pneumonectomy
* Home oxygen greater than 4L/minute
* Inability to adhere to assigned treatment prior to 48 hours of surgery or until transferred to a floor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Brainard, M.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- Unversity of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD

RESULTS

PARTICIPANT FLOW:
Groups:
- Heated Humidified High-flow Nasal Cannula (HHFNC) Oxygen: The intervention group received HHFNC O2 at a set flow of 40L/min. FiO2 was titrated by respiratory therapists to maintain SpO2 ≥ 90%. The HHFNC O2 apparatus included: 1) Air-Oxygen blender - capable of delivering 21-100% FiO2 at flow rates up to 60L/min, 2) Heated Humidifier - providing active heating and humidification to the delivered air-O2 blend, 3) Nasal cannula - larger diameter, slightly elongated nasal cannula with single limb connection to humidifier
  Heated humified high-flow nasal cannula Oxygen
- Standard Oxygen Therapy: The standard O2 treatment group received usual nasal cannula or face mask oxygen titrated by nurses as necessary to maintain SpO2 ≥ 90%.
  Standard oxygen therapy
Period: Overall Study
Arm/Group | Heated Humidified High-flow Nasal Cannula (HHFNC) Oxygen | Standard Oxygen Therapy
Started | 25 | 26
Completed | 18 | 26
Not Completed | 7 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Heated Humidified High-flow Nasal Cannula (HHFNC) Oxygen | Standard Oxygen Therapy | Total
Number analyzed (Participants) | 18 | 26 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 16 | 26
  >=65 years | 8 | 10 | 18
Age, Continuous [Mean (Full Range); unit: years] | 57 [18 to 100] | 59 [18 to 100] | 58 [18 to 100]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 8 | 14 | 22
Region of Enrollment [Number; unit: participants]
  United States | 18 | 26 | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Post-operative Pulmonary Complications
Description: The primary outcome "post-operative pulmonary complication" is defined as present if any one of the following criteria are met:
  * SpO2 < 90% with FiO2 ≥ 50%
  * Dyspnea at rest
  * Respiratory rate > 25 breaths/min
  * Active use of accessory respiratory muscles
  * PaO2/FiO2 ratio < 200
  * Escalation of therapy to non-invasive ventilation
  * Re-intubation
  * Occurrence of hospital-acquired pneumonia
  * Re-admission to the ICU
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Heated Humidified High-flow Nasal Cannula (HHFNC) Oxygen | Standard Oxygen Therapy
Number analyzed (Participants) | 18 | 26
Participants | 1 | 2
Statistical Analysis 1: Comparison: Heated Humidified High-flow Nasal Cannula (HHFNC) Oxygen vs Standard Oxygen Therapy; Test type: Other; p = 0.680, t-test, 1 sided

2. Secondary Outcome: Hospital Length of Stay
Description: length of stay from hospital admission to hospital discharge
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Heated Humidified High-flow Nasal Cannula (HHFNC) Oxygen | Standard Oxygen Therapy
Number analyzed (Participants) | 18 | 26
Days | 6.6 (2.1) | 9.5 (7)

3. Secondary Outcome: Lowest Oxygen Saturation Level Measured
Description: Lowest oxygen saturation level measured during hospitalization from admission to discharge
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | Heated Humidified High-flow Nasal Cannula (HHFNC) Oxygen | Standard Oxygen Therapy
Number analyzed (Participants) | 18 | 26
percentage of oxygen saturation | 88 (7) | 84 (7)

4. Secondary Outcome: ICU Length of Stay
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Heated Humidified High-flow Nasal Cannula (HHFNC) Oxygen | Standard Oxygen Therapy
Number analyzed (Participants) | 18 | 26
Days | 2 (1.2) | 3.2 (3.8)

ADVERSE EVENTS:
Arm/Group | Heated Humidified High-flow Nasal Cannula (HHFNC) Oxygen | Standard Oxygen Therapy
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/26
Other Adverse Events (participants affected / at risk) | 2/18 | 2/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Heated Humidified High-flow Nasal Cannula (HHFNC) Oxygen (N=18) | Standard Oxygen Therapy (N=26)
Pulmonary Complications (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No